CLINICAL TRIAL: NCT06697951
Title: Feasibility of Using Bubble Nasal Intermittent Pressure Ventilation Using the Neovent in Low-resource Settings
Brief Title: Feasibility of Using the Neovent in Low-Resource Settings
Acronym: Neovent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tina Slusher (Other)
Responsible Party: Sponsor-Investigator, Tina Slusher, MD, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-821
Record Dates: First submitted 2024-10-17; First posted 2024-11-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Distress of Newborn
Keywords: newborn; neonate; respiratory distress; Bilevel ventilation; low resource; Nepal; Nigeria
MeSH Terms: conditions — Pulmonary Atelectasis; Dyspnea

STUDY DESIGN:
Intervention Model Description: This is a study to test the usability of a low-cost way to do Non-invasive Positive Pressure Ventilation using the Neovent a device in lower resourced nurseries, Neovent has already be shown to be feasible in a higher resourced setting outside the United States in newborn infants with mild to moderate respiratory distress. The study plans to use the Neovent in lower-resourced nurseries who have respiratory distress in Nigeria and Nepal whose mothers give consent. The Neovent has been approved by regulatory bodies in India where the device is being manufactured for low-resource settings and will only be used for this study in Nigeria and Nepal and thus does not fall under FDA regulation. No patients will be enrolled from the United States therefore this study will not collect data for the purpose of approval for use in the United States.
Masking Description: Not possible to mask and not required for this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other): Newborns with mild to moderate respiratory distress whose caregivers give permission will be enrolled into the study
  Interventions: Device: bilevel ventilation with the Neovent

INTERVENTIONS:
Device: bilevel ventilation with the Neovent — Newborn infants with respiratory distress will be placed on the Neovent and we will see if study staff set up, use, and trouble shoot the Neovent correctly and see if study staff can monitor for safety problems in lower-resourced nurseries and to determine if the infants have any more problems than seen with bubble CPAP or Neovent in a higher resourced nursery including any more nasal irritation, abdominal distention, or clinically important amount of air around the lung (pneumothorax)

SUMMARY:
Breathing problems are a leading cause of newborn death/sickness worldwide but most of deaths are in low resources areas. Over 99% of newborn death is in countries with limited healthcare resources like Nigeria and Nepal.

Background For newborns who have trouble breathing, breathing with a machine that does not require an invasive breathing tube but only small nasal tubes is associated with lower rates of lung disease and less pneumonia or lung disease than newborns who have a breathing tube going into their lungs to help their breathing. Nasal Intermittent Positive Pressure Ventilation (NIPPV) is often used in high resource countries, but these machines are expensive. NIPPV gives many newborns the extra support needed to help with trouble breathing by providing extra pressure to help more air/oxygen get into their lungs. Neovent was designed to provide NIPPV at a much lower cost than machines than conventional machines. The Neovent has been shown to be safe and the device feasible in a higher resourced nursery than found in most nurseries in Nigeria and Nepal.

The primary and critical research gap this study will address is to show that investigators in lower resourced nurseries can use the Neovent thus demonstrating that this device is feasible to provide NIPPV for newborns with breathing problems without any more safety problems that those seen with the continuous positive airway pressure currently used in lower resourced nurseries in Nigeria and Nepal.

Aims The investigators believe NIPPV using the Neovent is feasible for use by healthcare providers in lower resourced nurseries in Nepal and Nigeria; that NIPPV provided by Neovent will be as safe as breathing support providing by machine CPAP and newborns on Neovent will not have more nasal irritation or nose bleeds, more stomach problems, or air around their lungs than newborns on machine CPAP.

Study design Newborns with mild-moderate breathing trouble whose mother/caregivers agrees will be placed on Neovent for 6 hours and monitored closely for any problems with the machine or newborn that are related to the machine especially injury to the nose, nosebleeds, swollen belly or abdomen, or air around the lungs.

Sample size We plan to enroll 70 newborn infants total from both sites in Nepal and Nigeria.

Next Steps The next step would be to do a study to determine if the Neovent is as good as other more expensive forms of breathing support for newborn infants.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION AND RATIONALE Infant respiratory distress is a leading cause of under-5 mortality worldwide, resulting in over one million infant deaths every year. Over 99% of these deaths occur in low to middle income countries For these vulnerable infants, noninvasive ventilation is preferred as it is associated with lower rates of chronic lung disease and ventilator-associated-pneumonia than invasive modes of ventilation. Widely used methods of noninvasive respiratory support for infants in respiratory distress include Nasal Continuous Positive Airway Pressure (NCPAP) and Nasal Intermittent Positive Pressure Ventilation (NIPPV). NCPAP consists of delivering a constant pressure, typically from 5 - 8 cm H2O, to recruit and stabilize the alveoli and improve ventilation and perfusion mismatch. NIPPV provides additional respiratory support with intermittent mandatory ventilation over the constant baseline pressure, e.g. 15 cm H2O over 5 cm H2O. The lower pressure is termed "P low" and the higher pressure is termed "P high". This additional respiratory support reduces the work of breathing3. In comparison with NCPAP, NIPPV has been shown to decrease the need for ventilation of preterm infants, decrease post-extubation failure and may further decrease the frequency of apneic episodes.

Bubble NCPAP is a simple, non-electric and easy to use means of delivering CPAP that has been successfully implemented across low and high resource settings 7,8. Unfortunately, until the present, there has not been an analogous simple, non-electric and easy to use means to deliver NIPPV. Conventional NIPPV equipment costs $10,000+, requires continuous electricity and requires many highly trained operators (physician, respiratory therapist, biomedical equipment technician), all of which serve as barriers to implementation in resource- constrained settings.

To address these barriers, a novel bubble NIPPV device, NeoVent, has been developed and shown to be both feasible and safe in a higher resourced nursery. With NeoVent, clinicians can independently set key parameters: upper level of pressure, lower level of pressure and rate (cycles/min). The technology is non-electric and visually intuitive to set up and operate. In the ASL 6000 infant lung simulator, NeoVent delivered comparable volumes and pressure waveforms as conventional ventilators. In sedated rabbits, NeoVent was able to achieve comparable ventilation, as demonstrated by arterial blood gas values, as a conventional ventilator13. In a first-in-human study of safety, NeoVent achieved a similar safety profile to bubble NCPAP 14. In a larger follow on study of safety, NeoVent again achieved a similar safety profile as bubble CPAP. Results have been published/presented in peer-reviewed forums including Pediatric Research, Respiratory Care, American Academy of Pediatrics, Indian Academy of Pediatrics, Canadian Society of Respiratory Therapists, Medicins Sans Frontieres and USAID/Gates Foundation's Grand Challenges in Global Health.

The investigators believe NIPPV using the Neovent is feasible for use by healthcare providers in lower resourced nurseries in Nepal and Nigeria; that NIPPV provided by Neovent will be as safe as breathing support providing by machine CPAP and newborns on Neovent will not have more nasal irritation or nose bleeds, more stomach problems, or air around their lungs than newborns on machine CPAP.

Primary Aim: Among infants (≤ 28 days) with respiratory distress settings, bubble NIPPV using the Neovent is feasible for use by healthcare providers in lower resourced nurseries in Nigeria and Nepal. This will test the hypothesis that at least 80% of healthcare providers' (clinicians/nurses) in lower resourced nurseries in Nigeria and Nepal can 1) set up, 2) operate and 3) troubleshoot bubble NIPPV using the Neovent and will be qualitatively assessed 3 months after introduction of the NIPPV in their NICU-based on survey/questionnaire/and demonstration.

Secondary Aims

* To demonstrate that health care providers in lower resourced nurseries in Nigeria and Nepal will be able evaluate for safety and correctly evaluate/stage nasal septal injury, nosebleeds, abdominal distention, clinically significant pneumothorax. This will test the hypothesis that healthcare providers in lower-resourced nurseries can correctly access for the primary safety concerns expected when using the Neovent.
* To demonstrate comparable rates of short-term complications (pneumothorax, nasal septal injury, nose bleeds, abdominal distention) between bubble NIPPV and those seen in previously with bubble CPAP. This will test the hypothesis that the side effects rates arse comparable in lower resourced nurseries to those seen both with bubble CPAP and with the Neovent in a higher resourced nurseries

Design: Over 6 months, 60 infants (≤28 days) and (≥30 weeks GA or ≥1000 grams if GA unknown) in mild to moderate respiratory distress in resource constrained referral hospitals in Nigeria and Nepal will be placed on bubble NIPPV with a Downes Score of 2-7. Health care providers (nurses together with physicians) ability to set up, operate and troubleshoot bubble NIPPV including monitoring for safety evaluating for nasal septal injury, abdominal distention and clinically significant pneumothorax will be qualitatively assessed.

Potential Impact: If bubble NIPPV is shown to be feasible and safe in resource constrained settings, this will justify further randomized controlled trials of efficacy.

Name and Description of Investigational Product or Intervention NeoVent delivers bubble Nasal Intermittent Positive Pressure Ventilation and is manufactured by Phoenix Medical Systems.

* 1 minute video describing device function: https://www.youtube.com/watch?v=cYZwbZK7lW4
* Product Description: https://www.phoenixmedicalsystems.com/infant-care/neovent Findings from Non-Clinical and Clinical Studies Pre-clinical studies In full-term and preterm neonatal manikins, bubble NIPPV reliably delivered alternating pressures consistent with standard NIPPV equipment9,10. In the IngMar ASL 5000 Test Lung simulator, delivered pressure waveforms and tidal volumes of bubble NIPPV were comparable with those of 2 conventional ventilators (Dräger Evita Infinity V500 and Hamilton G5) at the following pressure settings: 8/5, 12/5, and 15/5 cm H2O11,12. To simulate patients with pneumonia, transient tachypnea of the newborn and meconium aspiration syndrome, lung resistance was set at 100 cm H2O/L/s, and compliance set at 0.5, 1.0, and 2.0 mL/cm H2O15.

In anesthetized rabbits, bubble NIPPV reliably delivered two levels of airway pressure resulting in normalization of blood gases comparable to those achieved on a traditional ventilator13.

The delivery of comparable pressure waveforms and tidal volumes in lung simulators and normalization of arterial blood gas values in sedated animals suggests that bubble NIPPV provides treatment which may be comparable to traditional ventilator derived NIPPV. Thus, bubble NIPPV may provide clinicians in resource-limited settings with an additional, simple, non-electric treatment modality for the management of infant respiratory distress beyond bubble NCPAP alone.

Clinical studies Pilot data in a single center in Nepal In a cross-over cohort pilot in Nepal, 7 infants with moderate respiratory distress were randomized to 4 hours of treatment with bubble NCPAP vs bubble NIPPV followed by 4 hours of the alternate treatment. Vital signs, Downes' score (Retractions, Cyanosis, Respiratory Rate, Apnea, Expiratory Grunt) and O2 saturations were charted hourly. Survival and adverse events such as pneumothorax, nasal septal necrosis, necrotizing enterocolitis were recorded. All infants survived with similar median and interquartile values of vitals and Downes' scores, with no adverse events.

Safety in a single center in India At Paramitha Children's Hospital, a higher resourced nursery in Hyderabad, India, preterm (n=60) neonates with moderate respiratory distress were pragmatically allocated to bubble NCPAP (5-8 cm H2O) or bubble NIPPV (P high 8-10 cm H2O /P low 5-8 cm H2O) based on staff and equipment availability. Patient demographics on NCPAP and NIPPV were similar (mean +- SD; gestational age: 34.5 (1.4) vs. 34.6 (1.1) weeks; birth weight 2.2 (0.5) vs. 2.3 (0.4) kg; male: 67% vs. 67%) except for initial Respiratory Severity Score (RSS) which was 1.4 (0.4) on NCPAP vs. 2.4 (1.5) on NIPPV (p = .0008). Outcome measures included physiologic outcomes (hourly vital signs, Downes' score, FiO2), need for surfactant and need for intubation as well as complications including clinically relevant pneumothorax, septal necrosis, abdominal distention and other common complications of prematurity.

One patient in each arm developed minor nasal septal injury (grade 3 on NCPAP, grade 2 on NIPPV); no patients in either arm developed a clinically significant pneumothorax or abdominal distention. On NCPAP vs. NIPPV, 4 vs. 3 patients required a 1st dose of surfactant (excluding doses within the first two hours), and 1 vs. 0 patients required a second dose of surfactant. Two patients in the NCPAP arm required intubation in comparison with 4 patients in the NIPPV arm. There was a clinically and statistically significant improvement in FiO2 and Downes' score in NIPPV in comparison with NCPAP although patients on NIPPV did start with increased respiratory distress.

The similar rates of clinically significant nasal septal injury, pneumothorax and abdominal distention suggest that bubble NIPPV has a similar safety profile as bubble NCPAP for preterm infants in respiratory distress. Randomized controlled trials comparing the efficacy of bubble NCPAP and bubble NIPPV are warranted.

Given the demonstrated safety at one mid-resourced referral hospital, the investigators seek to study feasibility followed by efficacy in resource constrained hospitals.

Reference omitted but available upon request

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤ 28 days and > 30weeks and/or > 1000 gram (birthweight or admission weight if birthweight unknown)
* Mild to moderate respiratory distress (Downes' score 2 - 7)
* Parental/guardian permission (informed consent).

Exclusion Criteria:

* Congenital abnormality such that noninvasive positive pressure ventilation would be contraindicated (e.g. diaphragmatic hernia, cleft palate, tracheo-esophageal fistula)
* Need for immediate surgical intervention
* Suspected neuromuscular abnormality as evidenced by decreased tone
* Suspected cyanotic congenital cardiac disease or cardiac instability
* Severe life-threatening condition such that the doctor caring for the patient believes survival of patient will be less than 24 hours and/or parents request withdrawal of care

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Using Bubble Nasal Intermittent Pressure Ventilation Using the Neovent in Low-resource Settings | A physician will confirm the Neovent is set up properly within 1 hour after set up and will also confirm nurses' findings. Hourly fraction of inspired oxygen (FiO2), O2 saturation, respiratory rate, heart rate & Downes' score will be recorded for 6 hrs
  The investigators will measure the healthcare providers ability in lower-resource nurseries to 1) set up, 2) operate and 3) troubleshoot bubble NIPPV using the Neovent among infants (≤ 28 days) with respiratory distress.

SECONDARY OUTCOMES:
Healthcare assessment of safety | Infants will be assessed for clinically significant pneumothorax, septal necrosis, abdominal distention hourly and when the infant changes clinically and study physicians will verify the results are correct for 6 hrs
  The investigators will safety including the healthcare providers correct evaluation/staging of nasal septal injury, nosebleeds, abdominal distention, clinically significant pneumothorax and verify that the healthcares assessment is correct
Safety of Neovent | Infants will be assessed for clinically significant pneumothorax, septal necrosis, abdominal distention hourly and when the infant changes clinically and rates for 6 hrs infant in study and will be compared to the those from a higher resourced nursery
  Rates of clinically significant pneumothorax, nasal septal injury, nose bleeds, abdominal distention) will be measured and compared to those previously seen in between bubble NIPPV using the Neovent in lower resourced nurseries and those seen previously with bubble CPAP and Neovent in a higher resourced nursery

CONTACTS AND LOCATIONS:
Overall Officials: Tina M Slusher, MD, Principal Investigator — Hennepin Healthcare Research Institute; Isa Abulkadir, MBBS, Principal Investigator — Ahmadu Bellow University; Sunil John, MD, Principal Investigator — United Mission Hospital-Tansen, Nepal
Locations (2):
- United Mission Hospital-Tansen, Tānsen, Palpa District, Nepal
- Ahmadu Bello University, Zaria, Kano State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] John SC, Garg M, Muttineni M, Brearley AM, Rao P, Bhandari V, Slusher T, Murki S. Safety of bubble nasal intermittent positive pressure ventilation (NIPPV) versus bubble nasal continuous positive airway pressure (NCPAP) in preterm infants with respiratory distress. J Perinatol. 2024 Sep;44(9):1252-1257. doi: 10.1038/s41372-024-01904-8. Epub 2024 Feb 15. PMID 38361002
- [Background] Tsapis M, Mignot C, Katsahian S, Arbaoui H, Ayachi A. Case-control study of respiratory dynamic compliance in mechanically ventilated near-term newborns in a pre-hospital setting. Intensive Care Med. 2011 Dec;37(12):2008-14. doi: 10.1007/s00134-011-2377-z. Epub 2011 Oct 18. PMID 22005824
- [Background] John SC, Mohammed A, Church JT, John AV, Perkins EM, McLeod JS, Carr BD, Smith S, Barnett JH, Gustafson PA, Dick M, John SP. Bubble bilevel ventilation facilitates gas exchange in anesthetized rabbits. Pediatr Res. 2021 Feb;89(3):622-627. doi: 10.1038/s41390-020-0928-0. Epub 2020 May 1. PMID 32357365
- [Background] John SC, John AV, Moss AW, Gustafson PA, Fernando-Silva L, John SP. Bench Testing of a Bubble Noninvasive Ventilation Device in an Infant Lung Simulator. Respir Care. 2020 Sep;65(9):1339-1345. doi: 10.4187/respcare.07346. Epub 2020 Mar 24. PMID 32209707
- [Background] John SC, Barnett JD, Habben ND, Le HT, Cheng E, John SP, Gustafson PA. Development and Testing of a Bubble Bi-Level Positive Airway Pressure System. Respir Care. 2017 Sep;62(9):1131-1136. doi: 10.4187/respcare.05443. Epub 2017 May 30. PMID 28559463
- [Background] Martin S, Duke T, Davis P. Efficacy and safety of bubble CPAP in neonatal care in low and middle income countries: a systematic review. Arch Dis Child Fetal Neonatal Ed. 2014 Nov;99(6):F495-504. doi: 10.1136/archdischild-2013-305519. Epub 2014 Aug 1. PMID 25085942
- [Background] Lemyre B, Davis PG, de Paoli AG. Nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (NCPAP) for apnea of prematurity. Cochrane Database Syst Rev. 2002;(1):CD002272. doi: 10.1002/14651858.CD002272. PMID 11869635
- [Background] Lemyre B, Davis PG, De Paoli AG, Kirpalani H. Nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (NCPAP) for preterm neonates after extubation. Cochrane Database Syst Rev. 2017 Feb 1;2(2):CD003212. doi: 10.1002/14651858.CD003212.pub3. PMID 28146296
- [Background] Lemyre B, Laughon M, Bose C, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD005384. doi: 10.1002/14651858.CD005384.pub2. PMID 27976361
- [Background] Bhandari V. Nasal intermittent positive pressure ventilation in the newborn: review of literature and evidence-based guidelines. J Perinatol. 2010 Aug;30(8):505-12. doi: 10.1038/jp.2009.165. Epub 2009 Oct 22. PMID 19847188
- [Background] Schonherr U, Kuchle M, Handel A, Lang GK, Kuntze H, Naumann GO. ["Early" immunologic transplant reactions following perforating keratoplasty. A prospective clinical study]. Fortschr Ophthalmol. 1990;87(2):121-3. German. PMID 2358265
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534